CLINICAL TRIAL: NCT01305564
Title: A Prospective, Multi-Center Study of the Bard® Denali™ Retrievable Inferior Vena Cava Filter
Brief Title: A Prospective, Multi-Center Study of the Bard® Denali™ Retrievable Inferior Vena Cava Filter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-09-007
Record Dates: First submitted 2011-01-31; First posted 2011-02-28 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-02

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism (PE); Deep vein thrombosis (DVT); Vena cava; Vena cava filter; Inferior vena cava; Venous thromboembolic disease (VTED)
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Denali inferior vena cava filter (Experimental): All subjects enrolled will receive the Denali vena cava filter.
  Interventions: Device: Denali inferior vena cava filter

INTERVENTIONS:
Device: Denali inferior vena cava filter — The Denali inferior vena cava filter is a mechanical filtration device consisting of two levels of filtration (upper arms, lower legs), a retrieval hook to allow for retrieval using a standard snare, cranial and caudal anchors, and penetration limiters. The Denali filter is made from a laser cut nitinol tube.
  Other Names: DL900J; DL900F

SUMMARY:
The Bard® Denali™ Retrievable Inferior Vena Cava (IVC) study is a prospective, multi-center study which is intended to provide evidence of safety of the placement and retrieval of the Bard® Denali™ Retrievable Inferior Vena Cava Filter in subjects requiring IVC interruption to protect against pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* The subject or their legally authorized representative demonstrates understanding of the nature of the study and voluntarily provides written informed consent prior to any data collection or study procedures.
* The subject is ≥ 21 years old, must be either a male or non-pregnant female with an expected lifespan sufficient to allow for completion of all study procedures. A negative pregnancy test result (urine or blood) is required prior to implant. If an enrolled female becomes pregnant prior to study completion, participation in the study will be terminated.
* Based on Investigator judgment, the subject is at increased risk of PE requiring vena caval interruption. Note: Subjects diagnosed with acute DVT and/or PE must have objective confirmation based on imaging evidence of at least one of those diagnoses.
* Patients without PE or venous thromboembolic disease (VTED) who are at risk of PE may be enrolled in this trial. However, enrollment of these patients will be limited to a maximum of 40% of the total sample size.
* Based on Investigator's judgment, the subject has patent venous anatomy suitable for femoral or jugular/subclavian access for filter placement (e.g. no excessive tortuosity).
* The IVC is ≤ 28 mm in diameter at the intended implantation site based on radiographic imaging evidence.
* Based on Investigator's judgment, the filter can be safely placed such that the position of the filter tip is 1 cm below the lowest renal vein.
* Retrieval of the filter is expected within 180 days post placement. At the six month follow up, if the Investigator determines that the filter continues to be clinically indicated, the filter may be left in place until the risk of PE has passed or left in permanently. All patients not having their filter retrieved at six months will continue be followed to 24 months or one month post filter retrieval, whichever comes first.
* The subject has patent venous anatomy suitable for jugular access for retrieval of the filter based on imaging evidence within 48 hours prior to the filter placement procedure. Imaging mode will be at physician's discretion.
* The subject is willing to comply with the protocol requirements and specified follow-up evaluations.

Exclusion Criteria:

* The subject has a previously implanted filter in the IVC or superior vena cava (SVC).
* The subject has a duplicated or left-sided IVC.
* The subject has a severe spinal deformity that would impede access to the IVC for the filter placement or filter retrieval procedures.
* The subject has a serum creatinine ≥ 2 mg/dl (and not on dialysis) within seven days of study enrollment. Patients on dialysis are allowed to participate in this trial.
* The subject has a known uncorrectable bleeding diathesis or active coagulopathy.
* The subject has a life expectancy of < 25 months.
* The subject has a known allergy or sensitivity to nickel or titanium.
* The subject has a known allergy or sensitivity to iodinated contrast media, which cannot be adequately pre-medicated. NOTE: Alternative contrast agents are not permitted for the purposes of this study.
* The subject is currently participating in an investigational drug or another device study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Stavropoulos, MD, Principal Investigator — The Hospital of the University of Pennsylvania
Locations (22):
- United States (22):
  - University of Alabama Birmingham Medical Center, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Hartford Hospital, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Doctor's Hospital, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - HeartCare Midwest, Peoria, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - North Memorial Hospital, Robbinsdale, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denali Inferior Vena Cava Filter
Started | 200
Completed | 163
Not Completed | 37
Not completed — Death | 21
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: All subjects receiving a Denali vena cava filter.
Groups:
- Baseline Characteristics: All treated with Denali filter.
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (15.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 189
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 164
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Technical Success of Placement
Description: Technical success of filter placement is defined as the deployment of the filter such that the physician judges the location to be suitable to provide sufficient mechanical protection against Pulmonary Embolism.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Technical Success of Placement: Primary implant endpoint
Arm/Group | Technical Success of Placement
Number analyzed (Participants) | 200
percentage of participants | 99.5 [97.3 to 100]

2. Primary Outcome: Clinical Success of Placement
Description: Is the one-sided lower limit of the 95% confidence interval for the observed clinical success rate at least 80%? Clinical success of filter placement is defined as freedom from subsequent Pulmonary Embolism (PE), filter embolization, caval occlusion, filter and procedure related death, insertion adverse events (AEs), and technical failure of placement.
Time Frame: 6 months
Population: The denominator of 189 is equal to all of the subjects that completed the 6 month visit, had their filter retrieved, or experienced a component of the clinical success of placement endpoint regardless of follow-up duration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clinical Success of Placement
Number analyzed (Participants) | 189
percentage of participants | 95.2 [91.2 to 97.8]

3. Primary Outcome: Technical Success of Retrieval
Description: Technical success for retrieval is defined as retrieval of the filter such that the entire filter is retrieved intact.
Time Frame: 24 months
Population: The denominator of 124 is equal to the number of subjects that had a filter retrieval procedure (successful and unsuccessful retrievals). Subjects were not required to have a retrieval procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Technical Success of Retrieval
Number analyzed (Participants) | 124
percentage of participants | 97.6 [93.1 to 99.5]

4. Primary Outcome: Clinical Success of Retrieval
Description: Clinical success for retrieval is defined as successful technical retrieval of the filter without retrieval complications requiring intervention. Only the 121 successful retrievals are counted here.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clinical Success of Retrieval
Number analyzed (Participants) | 121
percentage of participants | 99.2 [95.5 to 100]

5. Secondary Outcome: Rate of Recurring Pulmonary Embolism
Description: Rate of recurrent Pulmonary Embolism while the filter is indwelling or one month post-retrieval.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Recurrent PE
Number analyzed (Participants) | 200
percentage of participants | 3.0 [1.1 to 6.4]

6. Secondary Outcome: Rate of New or Worsening Deep Vein Thrombosis
Description: Rate of new or worsening Deep Vein Thrombosis (DVT) from placement to the six month follow-up. Worsening DVT is defined as an extension of existing DVT to a new venous segment on ultrasound in patients that had DVT at the baseline visit.
Time Frame: 6 months
Population: The denominator of 188 is equal to the number of subjects completing the 6 month visit or with a filter retrieval procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | New or Worsening DVT
Number analyzed (Participants) | 188
percentage of participants | 10.1 [6.2 to 15.3]

7. Secondary Outcome: Filter Fracture
Description: Rate of filter fracture
Time Frame: 6 months
Population: The denominator of 186 is equal to the number of subjects that completed a 6 month follow-up or had their filter retrieved, with imaging completed to confirm lack of fracture.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filter Fracture
Number analyzed (Participants) | 186
percentage of participants | 0 [0.0 to 2.0]

8. Secondary Outcome: Filter Migration
Description: Rate of filter indwell complications of: migration >2cm.
Time Frame: 6 months
Population: The denominator of 186 is equal to the number of subjects that completed a 6 month follow-up or had their filter retrieved, with imaging completed to confirm lack of migration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filter Migration >2 cm
Number analyzed (Participants) | 186
percentage of participants | 0 [0.0 to 2.0]

9. Secondary Outcome: Filter Tilt at Placement
Description: Rate of filter indwell complications of: tilt >15°
Time Frame: Post-placement imaging
Population: Tilt was measured post-placement with vena cavagram.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filter Tilt: At Implant
Arm/Group | Filter Tilt
Number analyzed (Participants) | 200
percentage of participants | 0 [0.0 to 1.8]

10. Secondary Outcome: Filter Tilt at Retrieval
Description: Rate of filter indwell complications of: tilt >15°
Time Frame: Pre-retrieval imaging
Population: All patients undergoing a retrieval procedure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filter Tilt: At Retrieval
Arm/Group | Filter Tilt
Number analyzed (Participants) | 124
percentage of participants | 0 [0.0 to 2.9]

11. Secondary Outcome: Filter Penetration >3mm at Placement
Time Frame: Post-placement
Population: Penetration at Placement was measured immediately post-placement but prior to retrieval.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filter Penetration at Placement
Number analyzed (Participants) | 200
percentage of participants | 1.5 [0.3 to 4.3]

12. Secondary Outcome: Filter Penetration >3mm at Retrieval
Time Frame: Pre-retrieval
Population: The denominator of 124 is equal to the number of subjects undergoing a retrieval procedure with imaging to confirm penetration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filter Penetration at Retrieval
Number analyzed (Participants) | 124
percentage of participants | 1.6 [0.2 to 5.7]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the placement procedure and continued through the end of follow-up (24 months or 30-days post-retrieval).
Groups:
- Serious Adverse Events: Serious Adverse Events are reported for all 200 subjects and all serious events are reported.
  Non-serious adverse events are reported when the reported threshold for an event is at 5% or higher. This represents 175 subjects and not 200 for non-serious events.
Arm/Group | Serious Adverse Events
Serious Adverse Events (participants affected / at risk) | 90/200
Other Adverse Events (participants affected / at risk) | 138/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serious Adverse Events (N=200)
Anaemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis haemorrhagic (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 2
Catheter site haemorrhage (General disorders) | 1
Chest pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 3
Cholecystitis chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Acute graft versus host disease (Immune system disorders) | 1
Amyloidosis (Immune system disorders) | 1
Antiphospholipid syndrome (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 9
Sepsis (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 2
Breast cellulitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Extradural abscess (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Genitourinary tract infection (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Postoperative ileus (Injury, poisoning and procedural complications) | 2
Brain herniation (Injury, poisoning and procedural complications) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Open wound (Injury, poisoning and procedural complications) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Renal injury (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Vena cava injury (Injury, poisoning and procedural complications) | 1
Troponin increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastroesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Liposarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Urethral cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 3
Carpal tunnel syndrome (Nervous system disorders) | 1
Cervical cord compression (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Spinal claudication (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 3
Anuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 2
Pelvic haematoma (Reproductive system and breast disorders) | 1
Peyronie's disease (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 15
Hypotension (Vascular disorders) | 5
Arterial thrombosis (Vascular disorders) | 2
Shock haemorrhagic (Vascular disorders) | 2
Vena cava thrombosis (Vascular disorders) | 2
Venous thrombosis (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Superior vena caval stenosis (Vascular disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Factor V Leiden mutation (Congenital, familial and genetic disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Hernia (General disorders) | 1
Chest discomfort (General disorders) | 1
Clostridial Infection (Infections and infestations) | 1
Localized infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Viith nerve injury (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypovolemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metatstatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Esophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1
Facial palsy (Nervous system disorders) | 1
Piriformis syndrome (Nervous system disorders) | 1
Gynacomastia (Reproductive system and breast disorders) | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1
Skin hemorrhage (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Serious Adverse Events (N=200)
Nausea (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 18
Abdominal Pain (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 13
Back Pain (Musculoskeletal and connective tissue disorders) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 14
Urinary Tract Infection (Infections and infestations) | 18
Headache (Nervous system disorders) | 11
Anaemia (Blood and lymphatic system disorders) | 14
Tachycardia (Cardiac disorders) | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 12
Peripheral edema (General disorders) | 14
Pyrexia (General disorders) | 12
Deep Vein Thrombosis (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No